CLINICAL TRIAL: NCT04775758
Title: Atypical Orofacial Pain Diagnostics and Differentiation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Jan Pavel Rokicki, Administrator in Lithuanian University of Health Sciences Kaunas Clinics, Dentist, Oral Surgeon, Lithuanian University of Health Sciences
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-VZCH
Record Dates: First submitted 2021-02-21; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Persistent Idiopathic Facial Pain
Keywords: Persistent Idiopathic Facial Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atypical facial pain group (Experimental): Patients with clinally diagnosed G50.1 - atypical pain condition after all necessary diagnostic measures are taken to exclude a clear organic pathology (multiple diagnostic tests including MRI, CT and consultations from other specialists). Patients included in this study will undergo self-evaluating questionnaires and objective data analysis with facial expression analysis, galvanic skin response and heart rate. All tests are performed in one visit which will last up to an hour.
  Interventions: Behavioral: Self-evaluating questionnaires; Behavioral: iMotions analysis platform
- Maxillofacial fracture pain group (Active Comparator): Patients with maxillofacial fracture (S02.3, S02.4, S02.6.) will be subjected into control group. Patients included in this study will undergo self-evaluating questionnaires and objective data analysis with facial expression analysis, galvanic skin response and heart rate. All tests are performed in one visit which will last up to an hour.
  Interventions: Behavioral: Self-evaluating questionnaires; Behavioral: iMotions analysis platform

INTERVENTIONS:
Behavioral: Self-evaluating questionnaires — Patients are asked to describe their disease (gathering of anamnesis) and to categorize their symptoms according to their strength. Furthermore, patients complete self-evaluating questionnaires: Visual analog scale, Hospital anxiety and depression scale, Pittsburgh sleep quality index, Big five personality traits questionnaire.
Behavioral: iMotions analysis platform — While patients' anamnesis and questionnaire indexes are being gathered, iMotions software will gather facial expression analysis, galvanic skin response and heart rate data which will be compared with self-evaluating questionnaires.

SUMMARY:
Orofacial pain is diagnosed for more than 1.9 percent of general population and for 0.3 percent origin of the facial pain is unknown. Commonly atypical facial pain is treated as a neurological condition without an emotional or psychiatric evaluation. Since atypical pain and mood affective disorders can be related, patients do not receive proper care for this condition.

The aim of this study is to evaluate the relationship between atypical facial pain syndrome and affective mood disorders. We aim to assess patients' with no diagnosed organic pathology tendency towards anxiety, depression, sleep disorders and one of big five personality traits through self-rating questionnaires. We will compare the gathered data with biosensors from iMotions software.

ELIGIBILITY:
Experimental group The experimental group will consist only of adult patients (18-70years old), who were clinically diagnosed with atypical pain syndrome (G50.1) after all diagnostic measures were performed.

Inclusion criteria:

* Adult patients (18-70years old) who were clinically diagnosed with atypical pain syndrome (G50.1).
* Patients who accepted terms of this research and has signed informed consent form.
* Patients were not previously diagnosed with a psychiatric disorder.

Exclusion criteria:

* A potential participant of the study is not able to comprehend information regarding this study's protocol in both written and verbal forms or fails/refuses to sign an informed consent form.
* Patients who have a diagnosed organic pathology causing orofacial pain.
* Patients who are diagnosed with systemic diseases which may interfere with the study or patients who present with head or neck oncology pathologies.
* Patients who were previously diagnosed with a psychiatric disorder.

Control group Control group will consist of patients who were subjected to maxillofacial fracture (any jaw unilateral fracture). These patients will be involved in this study if they are hospitalized/or have visited Lithuanian University of Health Sciences hospital Kaunas Clinics Department of maxillofacial surgery.

Inclusion criteria:

* Adult patients (18-70year old) who have been diagnosed with orofacial pain due to jaw fracture (S02.3, S02.4, S02.6).
* Patients who have signed an informed consent form.
* Patients who were not previously diagnosed with a psychiatric disorder.

Exclusion criteria:

* A potential participant of the study is not able to comprehend information regarding this study's protocol in both written and verbal forms or fails/refuses to sign an informed consent form.
* Patients who are diagnosed with systemic diseases which may interfere with the study or patients who present with head or neck oncology pathologies.
* Patients who were previously diagnosed with a psychiatric disorder.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-02-27 (Estimated); Primary Completion 2021-07-22 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale | Assessment score gathered once (Day 1)
  Patients evaluate their spontaneous episodic pain before assessing self-evaluating questionnaires. Patient pain will be assessed using a visual analogue scale of 0-10, zero being no pain, ten being an unbearable/unimaginable pain. The higher score may lead to a possibilty of developing mood disorders.
Hospital anxiety and depression scale | Assessment score gathered once (Day 1)
  The Hospital anxiety and depression scale is a fourteen-item scale. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains. Patients were defined as having anxiety or depression or both if the score was 8 or more in the corresponding subscale.
Pittsburgh sleep quality index | Assessment score gathered once (Day 1)
  The Pittsburgh Sleep Quality Index contains 19 self-rated questions which measures seven aspects of sleep: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) habitual sleep efficiency, (5) sleep disturbances, (6) use of sleeping medication, and (7) daytime dysfunction. The 19 self-rated items are combined to form seven component scores, each of which has a range of 0-3 points (0 indicates no difficulty, while 3 indicates severe difficulty). The seven component scores are then summed to yield one global score, with a range of 0-21 points (0 indicating no difficulty, and 21 indicating severe difficulties in all the seven areas of sleep quality).
Big Five personality traits | Assessment score gathered once (Day 1)
  Big five personality traits questionnaire is a 25-item questionnaire compiled from Goldberg et al. 1999. Respondent chooses between a pair of adjectives and chooses an according score from one to seven. All personality dimensions are evaluated separately from specific pairs of adjectives and sum of these pairs scores. Lithuanian version is adapted from A.Bunevičius (2006).
Galvanic skin response. Valence | Assessment score gathered once (Day 1)
  Galvanic skin response peaks (countable) either total or within positive, negative and neutral condition valence.
Galvanic skin response. Amplitude | Assessment score gathered once (Day 1)
  Galvanic skin response is measured in microsiemens. Sudden rise in skin conductivity is called a peak. Peak amplitudes (in microsiemens) will be recorded and analysed. Average amplitude of peaks, either total or within positive, negative and neutral valence.
Galvanic skin response. Peaks/minute | Assessment score gathered once (Day 1)
  Peaks/minute (normalized measure) either total or within positive, negative and neutral valence.
Facial expression analysis. Duration of positive valence. | Assessment score gathered once (Day 1)
  Facial expression analysis determines the respondents' valence (negative, positive or neutral). The duration of positive valence (more than 30 percent threshold) will be assessed seconds.
Facial expression analysis. Duration of negative valence. | Assessment score gathered once (Day 1)
  Facial expression analysis determines the respondents' valence (negative, positive or neutral), the duration of negative valence (less than 30 percent threshold) will be assessed in seconds.
Facial expression analysis. Duration of neutral valence. | Assessment score gathered once (Day 1)
  Facial expression analysis determines the respondents' valence (negative, positive or neutral). The duration of neutral valence (from -30 percent to 30 percent threshold) will be assessed in seconds.
Facial expression analysis. Total duration. | Assessment score gathered once (Day 1)
  Facial expression analysis determines the respondents' valence (negative, positive or neutral). A total duration of the record (measuring time in seconds) will be used.

SECONDARY OUTCOMES:
Heart rate | Assessment score gathered once (Day 1)
  Using optical pulse sensors we aim to register beats per minute throughout the whole participation of the respondents.
Facial expression analysis (raw data) | Assessment score gathered once (Day 1)
  Average of probability scores for each emotion and facial expression.
Facial expression analysis threshold | Assessment score gathered once (Day 1)
  Fraction of time that an emotion or facial expression crosses the threshold of 30 percent.

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences Kaunas Clinics, Kaunas, Lithuania